CLINICAL TRIAL: NCT03091946
Title: Glycemic and Insulinemic Impact of Oats With Additional Dried Fruits, Nuts and Seeds Soaked Overnight in Skim Milk Versus Cream of Rice With Additional Dried Fruits, Nuts and Seeds
Brief Title: Glycemic and Insulinemic Impact of Oats With Additional Dried Fruits, Nuts and Seeds Soaked Overnight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1703
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Blood Glucose; Subjective Hunger, Insulin
Keywords: Oatmeal; Post-prandial glycemic response ; Post-prandial insulin response; Post-prandial hunger
MeSH Terms: conditions — Insulin Resistance | interventions — Nuts; Seeds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooked cream of rice (Placebo Comparator): Cream of rice with additional dried fruits, nuts and seeds cooked just prior to its consumption and served with skim milk as a beverage
  Interventions: Other: Cooked cream of rice with additional dried fruits, nuts and seeds
- Overnight oats (Experimental): Oats with additional dried fruits, nuts and seeds soaked overnight in skim milk
  Interventions: Other: Overnight oats with additional dried fruits, nuts and seeds

INTERVENTIONS:
Other: Overnight oats with additional dried fruits, nuts and seeds — Oatmeal
  Arms: Overnight oats
Other: Cooked cream of rice with additional dried fruits, nuts and seeds — Cooked cream of rice
  Arms: Cooked cream of rice

SUMMARY:
The purpose of this study is to compare the glucose, insulin and subjective hunger responses elicited by oats with additional dried fruits, nuts and seeds soaked overnight in skim milk and consumed cold versus Cream of Rice cereal with additional dried fruits, nuts and seeds cooked just prior to its consumption.

ELIGIBILITY:
Inclusion Criteria:

Male or non-pregnant females, 18-75 years of age, inclusive

* Body mass index (BMI) between 20.00 and 34.99 kg/m² inclusive at screening (visit 1).
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the Richardson Centre. Failure to comply will result in a rescheduled test visit.
* Normal fasting serum glucose (<6.3mmol/L).
* Willing to abstain from alcohol consumption for 24 h prior to all test visits.
* Willing to avoid vigorous physical activity for 24 h prior to all test visits.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Jones, the director of the Richardson Centre, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Known to be pregnant or lactating
* Unwillingness or inability to comply with the experimental procedures and to follow Richardson Centre safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at screening.
* Change in body weight of >3.5kg within 4 weeks of the screening visit.
* Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
* Exposure to any investigational drug product within 30 d prior to screening.
* Participation in any clinical trial 30 days prior to the start of this study.
* Participation in a PepsiCo clinical study in the past year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
incremental area under the blood glucose curve | 0-120 min
  The primary objective of this study is to compare the incremental area under the blood glucose curve from 0-120 min elicited by available carbohydrate matched portions of oats with additional dried fruits, nuts and seeds soaked overnight in skim milk and consumed cold versus Cream of Rice cereal with additional dried fruits, nuts and seeds.

SECONDARY OUTCOMES:
subjective hunger using Visual Analog Scale (VAS) | below baseline at 120, 180 and 240 min
  subjective hunger will be measured using VAS below baseline at 120, 180 and 240 min,
incremental areas under the curve (iAUC) of blood glucose | 0-180 min
  incremental areas under the curve (iAUC) of blood glucose from 0-180 min
iAUC of serum insulin | 0-120 min and 0-180 min
  iAUC of serum insulin from 0-120 min and 0-180 min

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Canada

IPD SHARING:
Plan to Share IPD: Undecided